CLINICAL TRIAL: NCT03567252
Title: Tanglewood to Table: A Walking Farmer's Market Group and Control
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dawn Brewer (Other)
Collaborators: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Responsible Party: Sponsor-Investigator, Dawn Brewer, Assistant Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 44215; P42ES007380 (NIH)
Record Dates: First submitted 2018-05-23; First posted 2018-06-25 (Actual); Results first posted 2021-07-23 (Actual); Last update posted 2021-07-23 (Actual); Status verified 2021-07

CONDITIONS: Dietary Habits
Keywords: Appalachia; Exercise
MeSH Terms: conditions — Feeding Behavior; Motor Activity

STUDY DESIGN:
Intervention Model Description: Participants will be compared between walking and non-walking groups to assess dietary behavior.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Walking Group (Experimental): Participants in this group will join an established walking group and travel by foot 1 kilometer to a local Farmer's Market. They will also receive handouts about nutrition information and nutritional choices.
  Interventions: Behavioral: Walking Group
- Non-Walking Group (No Intervention): Participants in this group will have no walking requirement. They will receive handouts about nutrition information and nutritional choices.

INTERVENTIONS:
Behavioral: Walking Group — Participants will walk 1 kilometer to a Farmer's Market.
  Arms: Walking Group

SUMMARY:
This program encourages community members to walk approximately 1 mile to the Whitesburg Farmers Market each Thursday or Saturday. The study aims to determine if walking to the market to receive vouchers improve health outcomes beyond controls who receive nutrition education.

DETAILED DESCRIPTION:
In the summer of 2018, community members of Whitesburg, Kentucky (KY) were recruited to join the Tanglewood to Table walking program, and community members of Harlan, KY were invited to serve as controls. Each Thursday or Saturday, participants report whether or not they walked the 1 mile trail to the farmers market, how many steps the walked in the previous 7 days and they reported which fruits and vegetables they consumed the previous week. The control group will receive nutrition education handouts. The program is from June 2018 - January 2019. Participants complete questionnaires about fruit and vegetable consumption and physical activity. Participants also provided physical and biological measurements. Recruiting for the 2018 Walking Program will begin in May.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years
* non-pregnant
* moderate to good health (able to walk approximately 1 mile)

Exclusion Criteria:

* under 18 years
* pregnant
* poor health (unable to walk approximately 1 mile)
* institutionalized adults
* impaired consent capacity
* prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 157 (Actual)
Dates: Start 2018-05-15 (Actual); Primary Completion 2019-05-21 (Actual); Study Completion 2019-05-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dawn Brewer, PhD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No
It depends on the quality of data.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 157 participants were enrolled. Of those, 90 participants were lost to follow-up or subsequently excluded based on protocol criteria. Sixty-seven participants (19 control and 48 intervention) engaged in the study.
Period: Overall Study
Arm/Group | Walking Group | Non-Walking Group
Started | 48 | 19
Completed | 48 | 19
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Walking Group | Non-Walking Group | Total
Number analyzed (Participants) | 48 | 19 | 67
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.8 (13.6) | 52.3 (11.4) | 50.5 (13.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 13 | 47
  Male | 14 | 6 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 43 | 14 | 57
  Unknown or Not Reported | 5 | 4 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 47 | 17 | 64
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 2
Region of Enrollment [Number; unit: participants]
  United States | 48 | 19 | 67

OUTCOME MEASURES:

1. Primary Outcome: Fruit Intake
Description: Participants will complete a survey indicating the total servings of fruit consumed (possible answers range from 1 serving in 3 months to 3 servings per day). Survey will be measured at baseline, 4 months, and 8 months. Data will be presented as average servings of fruit per group over time.
Time Frame: Baseline, 4 months and 8 months
Population: Not all participants were able to complete data collection for all three time points.
Measure: Mean (Standard Deviation); unit: servings of fruit per day
Arm/Group | Walking Group | Non-Walking Group
Number analyzed (Participants) | 48 | 15
servings of fruit per day
  baseline | 2.5 (2.9) | 2.9 (3.8)
  4 months (mid-point): number analyzed (Participants) | 48 | 13
  4 months (mid-point) | 2.3 (1.7) | 1.9 (1.6)
  8 months (post): number analyzed (Participants) | 48 | 11
  8 months (post) | 3.0 (4.2) | 1.6 (1.1)

2. Primary Outcome: Vegetable Intake
Description: Participants will complete a survey indicating the total servings of vegetables consumed (possible answers range from 1 serving in 3 months to 3 servings per day). Survey will be measured at baseline, 4 months, and 8 months. Data will be presented as average servings of vegetables per group over time.
Time Frame: Baseline, 4 months and 8 months
Population: Not all participants were able to complete data collection for all three time points.
Measure: Mean (Standard Deviation); unit: servings of vegetables per day
Arm/Group | Walking Group | Non-Walking Group
Number analyzed (Participants) | 48 | 16
servings of vegetables per day
  baseline: number analyzed (Participants) | 47 | 16
  baseline | 5.3 (5.1) | 2.6 (2.0)
  4 months (mid point): number analyzed (Participants) | 48 | 13
  4 months (mid point) | 5.8 (4.4) | 3.2 (2.1)
  8 months (post): number analyzed (Participants) | 48 | 11
  8 months (post) | 6.2 (7.9) | 2.6 (1.2)

3. Secondary Outcome: Change in Understanding of Plant-based Nutrients
Description: Participants will be asked a question demonstrating their understanding of the importance of ingesting plant-based nutrients at baseline, 4 months, and 8 months into the study. Possible answers are yes, no, or not sure. Data will be presented as the percent of participants in each group that understood the importance of plant-based nutrients over time.
Time Frame: Baseline, 4 months and 8 months
Population: Not all participants were able to complete data collection for all three time points.
Measure: Number; unit: percentage of participants
Arm/Group | Walking Group | Non-Walking Group
Number analyzed (Participants) | 47 | 15
percentage of participants
  baseline | 51.1 | 6.7
  4 months (mid-point): number analyzed (Participants) | 46 | 13
  4 months (mid-point) | 60.9 | 15.4
  8 months (post): number analyzed (Participants) | 45 | 11
  8 months (post) | 88.9 | 36.4

4. Secondary Outcome: Change in Believing in the Benefits of Plant-based Nutrients
Description: Participants will be asked a question demonstrating their appreciation of plant-based nutrients at baseline, 4 months, and 8 months into the study. Possible answers are yes, no, or not sure. Data will be presented as the percent of participants in each group that understood the importance of plant-based nutrients over time.
Time Frame: Baseline, 4 months and 8 months
Population: Not all participants were able to complete data collection for all three time points.
Measure: Number; unit: percentage of participants
Arm/Group | Walking Group | Non-Walking Group
Number analyzed (Participants) | 41 | 11
percentage of participants
  baseline: number analyzed (Participants) | 31 | 10
  baseline | 80.6 | 20.0
  4 months (mid-point) | 73.7 | 18.2
  8 months (post): number analyzed (Participants) | 41 | 8
  8 months (post) | 90.2 | 62.5

5. Secondary Outcome: Change in Believing in the Preventative Effects of Plant-based Nutrients
Description: Participants will be asked a question demonstrating their beliefs of plant-based nutrients at baseline, 4 months, and 8 months into the study. Possible answers are yes, no, or not sure. Data will be presented as the percent of participants in each group that understood the importance of plant-based nutrients over time.
Time Frame: Baseline, 4 months and 8 months
Population: Not all participants were able to complete data collection for all three time points.
Measure: Number; unit: percentage of participants
Arm/Group | Walking Group | Non-Walking Group
Number analyzed (Participants) | 41 | 11
percentage of participants
  baseline | 73.3 | 22.2
  4 months (mid-point): number analyzed (Participants) | 38 | 11
  4 months (mid-point) | 39.5 | 81.8
  8 months (post): number analyzed (Participants) | 41 | 8
  8 months (post) | 9.8 | 62.5

6. Secondary Outcome: Change in Believing in the Role of a Healthy Diet in Protecting Health From Pollutants
Description: Participants will be asked a question demonstrating their beliefs that a healthy diet might protect health from environmental pollutants at baseline, 4 months, and 8 months into the study. Possible answers are yes, no, or not sure. Data will be presented as the percent of participants in each group that understood the importance of a healthy diet over time.
Time Frame: Baseline, 4 months and 8 months
Population: Not all participants were able to complete data collection for all three time points.
Measure: Number; unit: percentage of participants
Arm/Group | Walking Group | Non-Walking Group
Number analyzed (Participants) | 48 | 19
percentage of participants
  baseline | 89.6 | 57.9
  4 months (mid-point): number analyzed (Participants) | 48 | 14
  4 months (mid-point) | 89.6 | 71.4
  8 months (post): number analyzed (Participants) | 47 | 11
  8 months (post) | 97.9 | 90.9

7. Secondary Outcome: Change in Knowledge of Which Foods Contain Phytonutrients
Description: Participants will be asked a question about which foods contain phytonutrients at baseline, 4 months, and 8 months into the study. Possible answers are meat, dairy, plant foods, all foods, or don't know. Data will be presented as the percent of participants in each group that correctly identified plant foods over time.
Time Frame: Baseline, 4 months and 8 months
Population: Not all participants were able to complete data collection for all three time points.
Measure: Number; unit: percentage of participants
Arm/Group | Walking Group | Non-Walking Group
Number analyzed (Participants) | 48 | 18
percentage of participants
  baseline | 56.3 | 22.2
  4 months (mid-point): number analyzed (Participants) | 47 | 14
  4 months (mid-point) | 59.6 | 21.4
  8 months (post): number analyzed (Participants) | 48 | 11
  8 months (post) | 77.1 | 45.5

8. Secondary Outcome: Change in Knowledge of Environmental Pollutants
Description: Participants will be asked to identify environmental pollutants from a list at baseline, 4 months, and 8 months into the study. Possible answers are polychlorinated biphenyls (PCBs), mercury, nitrites, all of those, none of those, or don't know. Data will be presented as the percent of participants in each group that correctly identified all of those over time.
Time Frame: Baseline, 4 months and 8 months
Population: Not all participants were able to complete data collection for all three time points.
Measure: Number; unit: percentage of participants
Arm/Group | Walking Group | Non-Walking Group
Number analyzed (Participants) | 48 | 19
percentage of participants
  baseline | 58.3 | 57.9
  4 months (mid-point): number analyzed (Participants) | 48 | 14
  4 months (mid-point) | 58.3 | 57.1
  8 months (post): number analyzed (Participants) | 48 | 11
  8 months (post) | 58.3 | 27.3

9. Secondary Outcome: Change in Days of Vigorous Exercise in the Last Week
Description: Participants will complete a survey at baseline, 4 months, and 8 months where they will be asked a number of days of the last 7 days that they participating in vigorous activity including the following: heavy lifting, digging, aerobics, or fast bicycling or other. Data will be presented as the average number of days of vigorous activity compared between groups over time
Time Frame: Baseline, 4 months and 8 months
Population: Not all participants were able to complete data collection for all three time points.
Measure: Mean (Standard Deviation); unit: days of vigorous exercise
Arm/Group | Walking Group | Non-Walking Group
Number analyzed (Participants) | 43 | 11
days of vigorous exercise
  baseline | 3.3 (2.1) | 4.2 (1.5)
  4 months (mid-point): number analyzed (Participants) | 43 | 10
  4 months (mid-point) | 2.7 (1.9) | 4.3 (1.7)
  8 months (post): number analyzed (Participants) | 30 | 5
  8 months (post) | 3.3 (1.7) | 3.0 (2.1)

10. Secondary Outcome: Change in Days of Moderate Exercise in the Last Week
Description: Participants will complete a survey at baseline, 4 months, and 8 months where they will be asked a number of days of the last 7 days that they participating in moderate activity including the following: light lifting, bicycling or other. Data will be presented as the average number of days of moderate activity compared between groups over time.
Time Frame: Baseline, 4 months and 8 months
Population: Not all participants were able to complete data collection for all three time points.
Measure: Mean (Standard Deviation); unit: days of moderate activity per week
Arm/Group | Walking Group | Non-Walking Group
Number analyzed (Participants) | 44 | 13
days of moderate activity per week
  baseline | 3.7 (2.2) | 3.7 (2.1)
  4 months (mid-point): number analyzed (Participants) | 44 | 9
  4 months (mid-point) | 3.7 (2.4) | 4.3 (1.3)
  8 months (post): number analyzed (Participants) | 34 | 8
  8 months (post) | 3.4 (1.7) | 2.9 (2.0)

11. Secondary Outcome: Change in Time Spent in Vigorous Exercise in the Last Week
Description: Participants will complete a survey at baseline, 4 months, and 8 months where they will be asked how much time in hours and minutes over the last 7 days that they participated in vigorous activity including the following: heavy lifting, digging, aerobics, or fast bicycling or other. Data will be presented as the average number of minutes or hours of vigorous activity compared between groups over time.
Time Frame: Baseline, 4 months and 8 months
Population: Not all participants were able to complete data collection for all three time points.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Walking Group | Non-Walking Group
Number analyzed (Participants) | 24 | 6
hours
  baseline | 2.4 (1.5) | 4.8 (4.4)
  4 months (mid-point): number analyzed (Participants) | 24 | 3
  4 months (mid-point) | 3.2 (2.5) | 4.0 (5.2)
  8 months (post): number analyzed (Participants) | 17 | 2
  8 months (post) | 2.9 (3.4) | 1.0 (1.4)

12. Secondary Outcome: Change in Time Spent in Moderate Exercise in the Last Week
Description: Participants will complete a survey at baseline, 4 months, and 8 months where they will be asked how much time in hours and minutes over the last 7 days that they participated in moderate activity including the following: lifting, bicycling or other. Data will be presented as the average number of minutes or hours of moderate activity compared between groups over time.
Time Frame: Baseline, 4 months and 8 months
Population: Not all participants were able to complete data collection for all three time points.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Walking Group | Non-Walking Group
Number analyzed (Participants) | 31 | 7
hours
  baseline | 2.6 (1.5) | 4.4 (2.8)
  4 months (mid-point): number analyzed (Participants) | 31 | 2
  4 months (mid-point) | 3.0 (2.9) | 1.0 (0)
  8 months (post): number analyzed (Participants) | 18 | 3
  8 months (post) | 2.7 (2.2) | 1.2 (1.0)

13. Secondary Outcome: Change in Time Spent Walking
Description: Participants will complete a survey at baseline, 4 months, and 8 months where they will be asked how many days over the last 7 days that they walked for at least 10 minutes. Data will be presented as the average number of minutes or hours of walking per day compared between groups over time.
Time Frame: Baseline, 4 months and 8 months
Population: Not all participants were able to complete data collection for all three time points.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Walking Group | Non-Walking Group
Number analyzed (Participants) | 28 | 7
hours
  baseline | 2.6 (2.2) | 4.1 (4.2)
  4 months (mid-point): number analyzed (Participants) | 27 | 5
  4 months (mid-point) | 2.7 (2.8) | 2.6 (2.1)
  8 months (post): number analyzed (Participants) | 25 | 3
  8 months (post) | 2.4 (2.1) | 1.0 (0)

14. Secondary Outcome: Change in Time Spent Sitting
Description: Participants will complete a survey at baseline, 4 months, and 8 months where they will be asked how many days over the last 7 days that they spent sitting. Data will be presented as the average number of minutes or hours of sitting per day compared between groups over time.
Time Frame: Baseline, 4 months and 8 months
Population: Not all participants were able to complete data collection for all three time points.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Walking Group | Non-Walking Group
Number analyzed (Participants) | 40 | 11
hours
  baseline | 4.8 (3.1) | 3.1 (1.2)
  4 months (mid-point): number analyzed (Participants) | 38 | 9
  4 months (mid-point) | 5.1 (3.6) | 4.7 (3.1)
  8 months (post): number analyzed (Participants) | 38 | 8
  8 months (post) | 5.0 (2.7) | 3.0 (2.3)

15. Secondary Outcome: Change in Dark Green Vegetable Consumption
Description: Participants will complete a survey at baseline, 4 months, and 8 months that will ask them if they eat at least 1.5 cups of dark green vegetables per week. Answers will include: 0= No, and I do not intend to in the next 6 months, 1= No, but I intend to in the next 6 months, 2= No, but I intend to in the next 30 days, 3=Yes, I have been but for less than 6 months, and 4=Yes I have been for the past 6 months. Data will be presented as the average intention to consume dark green vegetables compared between groups over time. Scores range from 0-4; higher scores indicate increased consumption.
Time Frame: Baseline, 4 months and 8 months
Population: Not all participants were able to complete data collection for all three time points.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Walking Group | Non-Walking Group
Number analyzed (Participants) | 48 | 18
score on a scale
  baseline | 3.0 (1.2) | 3.3 (1.3)
  4 months (mid-point): number analyzed (Participants) | 48 | 14
  4 months (mid-point) | 3.2 (1.0) | 3.1 (1.1)
  8 months (post): number analyzed (Participants) | 48 | 11
  8 months (post) | 3.3 (1.1) | 3.0 (1.2)

16. Secondary Outcome: Change in Red and Orange Vegetable Consumption
Description: Participants will complete a survey at baseline, 4 months, and 8 months that will ask them if they eat at least 5.5 cups of red and orange vegetables per week. Answers will include: 0=No, and I do not intend to in the next 6 months, 1=No, but I intend to in the next 6 months, 2=No, but I intend to in the next 30 days, 3=Yes, I have been but for less than 6 months, and 4=Yes I have been for the past 6 months. Data will be presented as the average intention to consume red and orange vegetables compared between groups over time. Scores range from 0-4; higher scores indicate increased consumption.
Time Frame: Baseline, 4 months and 8 months
Population: Not all participants were able to complete data collection for all three time points.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Walking Group | Non-Walking Group
Number analyzed (Participants) | 48 | 18
score on a scale
  baseline | 2.5 (1.2) | 2.4 (1.5)
  4 months (mid-point): number analyzed (Participants) | 48 | 14
  4 months (mid-point) | 2.7 (1.4) | 1.9 (1.3)
  8 months (post): number analyzed (Participants) | 48 | 11
  8 months (post) | 2.7 (1.4) | 2.6 (1.4)

17. Secondary Outcome: Change in Fruit and Vegetable Consumption
Description: Participants will complete a survey at baseline, 4 months, and 8 months that will ask them if they eat at least 5 cups of fruits and vegetables per week. Answers will include: 0=No, and I do not intend to in the next 6 months, 1=No, but I intend to in the next 6 months, 2=No, but I intend to in the next 30 days, 3=Yes, I have been but for less than 6 months, and 4=Yes I have been for the past 6 months. Data will be presented as the average intention to consume fruits and vegetables compared between groups over time. Scores range from 0-4; higher scores indicate increased consumption.
Time Frame: Baseline, 4 months and 8 months
Population: Not all participants were able to complete data collection for all three time points.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Walking Group | Non-Walking Group
Number analyzed (Participants) | 48 | 19
score on a scale
  baseline | 2.4 (1.2) | 2.5 (1.5)
  4 months (mid-point): number analyzed (Participants) | 48 | 14
  4 months (mid-point) | 2.9 (1.1) | 2.7 (1.2)
  8 months (post): number analyzed (Participants) | 48 | 11
  8 months (post) | 2.9 (1.2) | 2.4 (1.4)

18. Secondary Outcome: Change in Fruit Consumption
Description: Participants will complete a survey at baseline, 4 months, and 8 months that will ask them if they eat at least 2 cups of fruits per week. Answers will include: 0= No, and I do not intend to in the next 6 months, 1=No, but I intend to in the next 6 months, 2=No, but I intend to in the next 30 days, Y3=es, I have been but for less than 6 months, and 4=Yes I have been for the past 6 months. Data will be presented as the average intention to consume fruits compared between groups over time. Scores range from 0-4; higher scores indicate increased consumption.
Time Frame: Baseline, 4 months and 8 months
Population: Not all participants were able to complete data collection for all three time points.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Walking Group | Non-Walking Group
Number analyzed (Participants) | 48 | 19
score on a scale
  baseline | 2.4 (1.3) | 2.0 (1.6)
  4 months (mid-point): number analyzed (Participants) | 48 | 14
  4 months (mid-point) | 2.4 (1.3) | 2.4 (0.9)
  8 months (post): number analyzed (Participants) | 48 | 11
  8 months (post) | 2.6 (1.2) | 2.5 (1.3)

19. Secondary Outcome: Change in Walking 1 Mile Per Day
Description: Participants will complete a survey at baseline, 4 months, and 8 months that will ask them if they walk at least 1 mile per day. Answers will include:0=No, and I do not intend to in the next 6 months, 1=No, but I intend to in the next 6 months, 2=No, but I intend to in the next 30 days, 3=Yes, I have been but for less than 6 months, and 4= Yes I have been for the past 6 months. Data will be presented as the average intention to walk 1 mile per day compared between groups over time. Scores range from 0-4; higher scores indicate increased walking.
Time Frame: Baseline, 4 months and 8 months
Population: Not all participants were able to complete data collection for all three time points.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Walking Group | Non-Walking Group
Number analyzed (Participants) | 47 | 18
score on a scale
  baseline | 2.9 (1.2) | 3.1 (1.4)
  4 months (mid-point): number analyzed (Participants) | 47 | 14
  4 months (mid-point) | 3.4 (0.9) | 2.6 (1.3)
  8 months (post): number analyzed (Participants) | 47 | 11
  8 months (post) | 3.4 (1.0) | 1.9 (1.5)

20. Secondary Outcome: Change in Leisure Time and Physical Activity
Description: Participants will complete a survey at baseline, 4 months, and 8 months that will ask them if they get about 30 minutes of leisure time/recreational physical activity or exercise every day. Answers will include: 0= No, and I do not intend to in the next 6 months, 1=No, but I intend to in the next 6 months, 2=No, but I intend to in the next 30 days, 3=Yes, I have been but for less than 6 months, and 4=Yes I have been for the past 6 months. Data will be presented as the average intention to get 30 minutes of exercise every day compared between groups over time. Scores range from 0-4; higher scores indicate increased activity.
Time Frame: Baseline, 4 months and 8 months
Population: Not all participants were able to complete data collection for all three time points.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Walking Group | Non-Walking Group
Number analyzed (Participants) | 48 | 18
score on a scale
  baseline | 3.1 (1.1) | 2.9 (1.4)
  4 months (mid-point): number analyzed (Participants) | 48 | 14
  4 months (mid-point) | 3.3 (0.8) | 2.8 (1.1)
  8 months (mid-point): number analyzed (Participants) | 48 | 11
  8 months (mid-point) | 3.3 (1.0) | 2.6 (1.4)

21. Secondary Outcome: Change in General Health
Description: Participants will complete a survey at baseline, 4 months, and 8 months that will ask them to state if they consider their health to be: 0=poor, 1=fair, 2=good, 3=very good, or 4=excellent. Data will be presented as the average ranking of individual health compared between groups over time. Scores range from 0-4; higher scores indicate a higher perception of health.
Time Frame: Baseline, 4 months and 8 months
Population: Not all participants were able to complete data collection for all three time points.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Walking Group | Non-Walking Group
Number analyzed (Participants) | 48 | 19
score on a scale
  baseline | 1.8 (0.9) | 2.1 (0.9)
  4 months (mid-point): number analyzed (Participants) | 47 | 14
  4 months (mid-point) | 2.0 (0.9) | 1.7 (1.0)
  8 months (post): number analyzed (Participants) | 47 | 11
  8 months (post) | 2.1 (1.0) | 1.8 (1.3)

22. Secondary Outcome: Change in Participation in Program
Description: Participants will complete a survey at baseline, 4 months, and 8 months that will ask them why they decided to participate in the program. Data will be presented as the number of participants that selected the most frequent answer ("to receive a farmer's market voucher").
Time Frame: Baseline, 4 months and 8 months
Population: Not all participants were able to complete data collection for all three time points. Participants in the control group were not asked to respond to this question.
Measure: Count of Participants; unit: Participants
Arm/Group | Walking Group | Non-Walking Group
Number analyzed (Participants) | 47 | 0
Participants
  baseline | 19 |
  4 months (mid-point): number analyzed (Participants) | 44 | 0
  4 months (mid-point) | 18 |
  8 months (post) | 24 |

23. Other Pre Specified Outcome: Change in Total Steps Taken Per Day
Description: Participants in the walking group will be issued pedometers to measure the total number of steps taken per day. Data will be collected weekly for the duration of the study. Data presented as the average number of steps per day.
Time Frame: Baseline, 4 months and 8 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse event data were not collected for this study.
Description: Serious adverse event, non-serious adverse event, and mortality data were not collected for this study.
Arm/Group | Walking Group | Non-Walking Group
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-05-14): https://cdn.clinicaltrials.gov/large-docs/52/NCT03567252/Prot_SAP_001.pdf
  • Informed Consent Form (2018-07-31): https://cdn.clinicaltrials.gov/large-docs/52/NCT03567252/ICF_000.pdf